CLINICAL TRIAL: NCT02919969
Title: A Multicenter Phase 2 Clinical Trial of Pembrolizumab in Metastatic Anal Cancer
Brief Title: Pembrolizumab in Metastatic Anal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, James Cleary, MD, PhD, MD/PhD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-301
Record Dates: First submitted 2016-09-02; First posted 2016-09-30 (Estimated); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Anal Cancer
Keywords: Anal Cancer
MeSH Terms: conditions — Anus Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): * Pembrolizumab is administered every 3 week intravenously
  * Dosage to be determine by physician
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
  Other Names: Keytruda; MK-3475

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for advanced anal cancer.

The following intervention will be involved in this study:

-Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for Advanced Anal Cancer, but it has been approved for other uses.

Pembrolizumab, also known as KEYTRUDA or MK-3475, is approved in the USA and several other countries to treat a type of skin cancer called Malignant Melanoma.

In this research study the investigators are studying an investigational drug called Pembrolizumab, which is a monoclonal antibody. Monoclonal antibodies are manmade and mimic proteins in the immune system by attaching to specific proteins in the body. T cells are cells in the immune system that are controlled by PD-1. PD-1 is a protein on the T cells that prevent the body from overproducing T cells. Pembrolizumab targets PD-1, attaches to it and blocks its action. By preventing PD-1 from working, T cell production rises and the body's immune system may increase its action against Cancer cells. Clinical and laboratory studies using pembrolizumab suggest that pembrolizumab may be useful in shrinking certain tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have metastatic anal cancer that has been histologically confirmed.
* There is no limit to the number of prior therapies.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function, all screening labs must be performed within 10 days of treatment initiation.

Adequate Organ Function Laboratory Values

System Laboratory Value

* Hematological

  * Absolute neutrophil count (ANC) ≥1,500 /mcL
  * Platelets ≥80,000 / mcL
  * Hemoglobin ≥8.5 g/dL or ≥5.6 mmol/L
* Renal

  --Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Hepatic

  * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
  * Albumin >2.8 mg/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Creatinine clearance should be calculated per institutional standard.
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 7.4). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Subjects requiring systemic steroids are excluded from the trial. The use of physiologic doses of corticosteroids may be approved after discussion with the sponsor.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: Subjects with ≤ Grade 2 neuropathy and alopecia are an exception to this criterion and may qualify for the study.
  * Note: If subject received major surgery, they must wait ≥ 3 weeks prior to starting study treatment. They must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has an active infection requiring systemic therapy.
* Patients that require supplemental oxygen are excluded.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* HIV+ positive patients are eligible if their CD4+ count ≥ 300/μL and they have an undetectable viral load. In addition, they must be currently receiving Highly Active Antiretroviral Therapy (HAART) and be under the care of an Infectious Diseases specialist.
* Patients with hepatitis B and hepatitis C must be under the care of viral hepatitis expert consultant. Patients with hepatitis B are required to be treated with anti-HBV treatment (e.g., entecavir). Patients with hepatitis C need to have received prior and/or ongoing hepatitis C treatment.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2023-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Cleary, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients were consented and screened for the trial
Pre-assignment Details: 32 patients met eligibility criteria and were treated with the study drug
Groups:
- Pembrolizumab: Pembrolizumab is administered every 3 week intravenously. Dosage to be determined by physician
  Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 32
Completed | 1
Not Completed | 31
Not completed — Lack of Efficacy | 22
Not completed — Death | 4
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients who met eligibility
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 60.9 [36 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate of pembrolizumab in metastatic anal cancer patients will be evaluated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions. A complete response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Disease was evaluated radiologically at baseline and every 3 cycles on treatment. The median follow-up was 12.6 months. All registered patients received at least one infusion of pembrolizumab and were treated for a median of 2 months (range: 0-23 months)
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
probability | 11.1 [2.4 to 29.2]

2. Secondary Outcome: PD-L1 Positive Response Rate
Description: Response rate in PD-L1 positive metastatic anal cancer patients will be evaluated by RECIST 1.1.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
probability | 13.0 [3.99 to 35.1]

3. Secondary Outcome: Overall Survival
Description: Evaluate the durability of pembrolizumab responses in PD-L1 positive metastatic anal cancer patients by measuring median overall survival.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
months | 13.6 [6.5 to 17.7]

4. Secondary Outcome: Progression Free Survival
Description: Evaluate the durability of pembrolizumab responses in PD-L1 positive metastatic anal cancer patients by measuring median progression free survival.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
months | 2.2 [1.9 to 4.1]

5. Secondary Outcome: Incidence of Adverse Events to Evaluate the Safety and Tolerability of Pembrolizumab
Description: Assess how well pembrolizumab is tolerated in patients with metastatic anal cancer by evaluating adverse events by CTCAE v4.0. Safety was assessed every 3 Weeks, from the time the informed consent is signed through 90 days following cessation of treatment. The median follow-up period was 12.6 months (range= 0.6-51.6 months).
Time Frame: Every 3 Weeks, from the time the informed consent is signed through 90 days following cessation of treatment "Every 3 Weeks, from the time the informed consent is signed through 30 days following cessation of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Pembrolizumab: * Pembrolizumab is administered every 3 week intravenously
  * Dosage to be determine by physician
  Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 32
Participants | 25

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the time the consent form was signed every 3 weeks from the time the informed consent is signed through 90 days following cessation of treatment. The median follow-up period was 12.6 months (range= 0.6-51.6 months).
Description: A serious adverse event was any adverse event occurring at any dose or during any use of pembrolizumab that:
  * Results in death;
  * Is life threatening;
  * Results in persistent or significant disability/incapacity;
  * Results in or prolongs an existing inpatient hospitalization;
  * Is a congenital anomaly/birth defect;
  * Is a new cancer (that is not a condition of the study);
  * Is associated with an overdose;
  * Is another important medical event
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 24/32
Serious Adverse Events (participants affected / at risk) | 13/32
Other Adverse Events (participants affected / at risk) | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab (N=32)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Colitis (Gastrointestinal disorders) | 1
Sudden death NOS (General disorders) | 2
Syncope (Nervous system disorders) | 1
Infections and Infestations (Infections and infestations) | 1 — Infection
Urinary tract Obstruction (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Hydronephrosis
Creatinine increased (Investigations) | 1
Hypertension (Vascular disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 — C. Diff
Scrotal pain (Reproductive system and breast disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=32)
Alanine aminotransferase increased (Investigations) | 2 (4)
Alkaline phosphatase increased (Investigations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 6 (8)
Blood bilirubin increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (2)
Fatigue (General disorders) | 11 (12)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 4 (4)
Localized edema (General disorders) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Neutrophil count decreased (Investigations) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (10)
Skin/subcutaneous tissue disorders; Other, specify (mouth sore) (Skin and subcutaneous tissue disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02919969/Prot_SAP_000.pdf